CLINICAL TRIAL: NCT01073124
Title: Sensitivity of the Saline Load Test With and Without Methylene Blue Dye in the Diagnosis of Traumatic Knee Arthrotomies
Brief Title: Sensitivity Diagnosing Traumatic Knee Injuries With and Without Injection of Blue Dye Into the Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NMCSD.2008.0006
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Traumatic Knee Arthrotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Active Comparator): Normal Saline injected intraarticularly into the knee joint
  Interventions: Procedure: Saline Load Test
- Dilute Methylene Blue Dye (Experimental): 1 ml methylene blue dye per 500 ml normal saline injected intraarticularly into the knee
  Interventions: Procedure: Saline Load Test

INTERVENTIONS:
Procedure: Saline Load Test — Intraarticular injection of dilute methylene blue dye (1 ml per 500 ml normal saline) or normal saline into the knee joint through a lateral suprapatellar injection site. Maximum injection of 180 ml.

SUMMARY:
The purpose of this study is to determine if adding blue dye improves the saline load test, which is a way to detect a traumatic intraarticular knee injury by injecting normal saline into the knee and looking for outflow through the wound.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with diagnosis warranting elective knee arthroscopy

Exclusion Criteria:

* Pregnant women
* Decreased knee range of motion (flex < 125, ext <0)
* Active infection of knee joint
* history of or current intraarticular knee malignancy
* history of open traumatic injury of the knee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Volume (mm) injected at time of outflow | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Metzger, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No